CLINICAL TRIAL: NCT04465370
Title: A Prospective, Single-Arm, Nonrandomized, Observational Study of Cardiac Output Monitoring in Pediatric Patients
Brief Title: Pediatric Cardiac Output Monitoring Observational Study
Acronym: POGO
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-08
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Results first posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-09

CONDITIONS: Pediatric ALL
Keywords: Hemodynamic Monitoring; Cardiac Output
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: Hemosphere Advanced Monitoring System, ClearSight 1.5, Swan-Ganz Catheter, Flotrac, Foresight — A Swan-Ganz catheter, FloTrac transducer, ClearSight finger cuff and ForeSight Elite sensors will be placed prior to the start of the catheterization procedure. Intermittent cardiac output and other hemodynamic parameters will be collected throughout the duration of the procedure and analyzed according to the Statistical Analysis Plan.

SUMMARY:
To assess Cardiac Output Monitoring in pediatric subjects by comparing FloTrac and ClearSight system to intermittent thermodilution Swan-Ganz, in order to expand the indications of FloTrac, ClearSight and Swan-Ganz thermodilution pulmonary artery catheter to the pediatric population 12 to 18 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 12 to 18 years of age
* Subjects who have signed the Informed Consent Form
* Subjects who are projected to receive Swan-Ganz catheter as part of procedure/standard of care with intermittent cardiac output measures
* For those Subjects who have had a cardiac transplant,Subjects who are at least 2 weeks post cardiac transplantation
* Subjects with planned pressure monitoring with an arterial line

Exclusion Criteria:

* Subjects with contraindications for Pulmonary Artery Catheters Placement and monitoring (recurrent sepsis, or with hypercoagulopathy);
* Subjects with contraindications for Arterial Line Placement;
* Subjects with an extreme contraction of the smooth muscle in the arteries and arterioles in the lower arm and hand (i.e., Raynaud's Disease).
* Subjects with a physical site area too limited for proper Sensor placement
* Subjects with finger size less than the smallest finger cuff size
* Documented ≥ moderate pulmonary hypertension (PAPm > 25mmHg, PVRI > 3.0 WUxm2)
* Presence of intracardiac shunting (i.e., ASD, VSD)
* Aorto-pulmonary collaterals
* ≥ Moderate tricuspid regurgitation, per echocardiogram criteria
* > Moderate Aortic or pulmonary regurgitation, per echocardiogram criteria
* Persistent cardiac arrythmias during the cardiac catheterization period (> 3min)
* Vascular abnormalities of the arterial system (i.e., connective tissue disorders, mid-aortic syndrome)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Males and Females, 12 to 18 years of age at the time of screening. Who presenting to Cardiac Catheterization Lab for right heart catheterizations.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UF Health Shands Children's Hospital, Gainesville, Florida
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were a total of 89 subjects enrolled. After applying the pre-determined rejection criteria for hemodynamic instability or poor signal quality, there were 60 Evaluable Pivotal Subjects.
Groups:
- Device: Hemosphere Advanced Monitoring System, ClearSight, Swan-Ganz Catheter, Flotrac, Foresight: A Swan-Ganz catheter, FloTrac transducer, ClearSight finger cuff and ForeSight Elite sensors will be placed prior to the start of the catheterization procedure. Intermittent cardiac output and other hemodynamic parameters will be collected throughout the duration of the procedure and analyzed according to the Statistical Analysis Plan.
Period: Overall Study
Arm/Group | Device: Hemosphere Advanced Monitoring System, ClearSight, Swan-Ganz Catheter, Flotrac, Foresight
Started | 89
Completed | 60
Not Completed | 29

BASELINE CHARACTERISTICS:
Arm/Group | Device: Hemosphere Advanced Monitoring System, ClearSight, Swan-Ganz Catheter, Flotrac, Foresight
Number analyzed (Participants) | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 89
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.3 (1.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 21
  White | 60
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Bias of FloTrac Arterial Pressure Cardiac Output (L/Min) Against Swan Ganz Invasive Cardiac Output
Description: Bias of FloTrac Arterial Pressure Cardiac Output (APCO) against Swan Ganz Invasive Cardiac Output (ICO) was calculated via Bland-Altman analysis
Time Frame: Duration of cardiac catheterization procedure, an average of 2 hours
Population: After applying the pre-determined data exclusion criteria for hemodynamic instability or poor signal quality, there were 60 Evaluable Pivotal Subjects in each of the comparison groups.
Measure: Mean (95% Confidence Interval); unit: L/min
Groups:
- Swan-Ganz ICO vs. FloTrac CO - Bias: Group of pediatric subjects aged 12-18 comparing Swan-Ganz intermittent CO [SG-ICO] to FloTrac CO [FTCO].
Arm/Group | Swan-Ganz ICO vs. FloTrac CO - Bias
Number analyzed (Participants) | 60
L/min | 0.49 [0.30 to 0.68]

2. Primary Outcome: Precision of FloTrac Arterial Pressure Cardiac Output (L/Min) Against Swan Ganz Invasive Cardiac Output
Description: Precision of FloTrac Arterial Pressure Cardiac Output (APCO) against Swan Ganz Invasive Cardiac Output (ICO) was calculated via Bland-Altman analysis
Time Frame: Duration of cardiac catheterization procedure, an average of 2 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Groups:
- Swan-Gan ICO vs. FloTrac CO - Precision: Group of pediatric subjects aged 12-18 comparing Swan-Ganz intermittent CO [SG-ICO] to FloTrac CO [FTCO].
Arm/Group | Swan-Gan ICO vs. FloTrac CO - Precision
Number analyzed (Participants) | 60
L/min | 1.11 [0.92 to 1.30]

3. Primary Outcome: Bias of ClearSight Arterial Pressure Cardiac Output (L/Min) Against Swan Ganz Invasive Cardiac Output
Description: Bias of ClearSight Arterial Pressure Cardiac Output (APCO) against Swan Ganz Invasive Cardiac Output (ICO) was calculated via Bland-Altman analysis
Time Frame: Duration of cardiac catheterization procedure, an average of 2 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Groups:
- Swan-Ganz ICO vs. ClearSight CO - Bias: Group of pediatric subjects aged 12-18 comparing Swan-Ganz intermittent CO [SG-ICO] to ClearSight CO [CSCO].
Arm/Group | Swan-Ganz ICO vs. ClearSight CO - Bias
Number analyzed (Participants) | 60
L/min | 0.41 [0.21 to 0.61]

4. Primary Outcome: Precision of ClearSight Arterial Pressure Cardiac Output (L/Min) Against Swan Ganz Invasive Cardiac Output
Description: Precision of ClearSight Arterial Pressure Cardiac Output (APCO) against Swan Ganz Invasive Cardiac Output (ICO) was calculated via Bland-Altman analysis
Time Frame: Duration of cardiac catheterization procedure, an average of 2 hours
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: L/min
Groups:
- Swan-Ganz ICO vs. ClearSight CO - Precision: Group of pediatric subjects aged 12-18 comparing Swan-Ganz intermittent CO [SG-ICO] to ClearSight CO [CSCO].
Arm/Group | Swan-Ganz ICO vs. ClearSight CO - Precision
Number analyzed (Participants) | 60
L/min | 1.11 [0.92 to 1.30]

ADVERSE EVENTS:
Time Frame: Duration of the procedure through 30 days after procedure, plus or minus 14 days
Groups:
- Treatment Population: All subjects were provided with Swan-Ganz, FloTrac, and ClearSight monitors.
Arm/Group | Treatment Population
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 5/89
Other Adverse Events (participants affected / at risk) | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Population (N=89)
Admission For Atg Treatment For Rejection (Cardiac disorders) | 1 (1)
Transplant Rejection Amr Grade 2 (Cardiac disorders) | 1 (1)
Cardiac (General disorders) | 1 (1)
Other (Immune system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT04465370/Prot_SAP_000.pdf